CLINICAL TRIAL: NCT02253069
Title: A Study of Polyhexanide-based Antiseptic in Full-thickness Surgical Wounds in Dermatologic Surgery
Brief Title: PHMB-based Antiseptic Use in Full-thickness Surgical Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Vinnova (Other Government)
Responsible Party: Principal Investigator, Karim Saleh, Dr., Region Skane
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Regionskane
Record Dates: First submitted 2014-09-24; First posted 2014-10-01 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Surgical Site Infections
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PHMB-based antiseptic (Experimental): Applying Prontosan antiseptic solution to tie-over dressings
  Interventions: Device: Applying Prontosan antiseptic solution to tie-over dressings
- Control (Placebo Comparator): Applying water to tie-over dressings
  Interventions: Device: Applying Placebo to tie-over dressings

INTERVENTIONS:
Device: Applying Prontosan antiseptic solution to tie-over dressings — Applying a PHMB-based antiseptic to tie-over dressings
  Arms: PHMB-based antiseptic
Device: Applying Placebo to tie-over dressings — Placebo control
  Arms: Control

SUMMARY:
To study the effect of applying a PHMB-based antiseptic solution to tie-over dressings in full-thickness surgical wounds in dermatologic surgery in order to minimise the development of surgical site infections. The bacterial dynamics in wounds pre-,intra-, and postoperatively will be examined in order to understand the pathogenesis of surgical site infections better.

DETAILED DESCRIPTION:
40 patients with suspected skin cancer in the face planned for full-thickness surgery will be randomised into two groups: One will receive a traditional tie-over dressing saturated with NaCl and the other group will receive a tie-over dressing saturated with a PHMB-based antiseptic. A quantitative and qualitative bacterial analysis of wounds by using a modified Levine's swabbing technique will be carried out pre-,intra-,and postoperatively. The effect of nasal colonisation with S.aureus on the development of surgical site infections will be investigated. All wounds will be followed a week after surgery to assess development of infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for full-thickness skin grafting in the face

Exclusion Criteria:

* Patients with no diabetes
* Patients with no current/previous/recent antibiotic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Measuring colony forming units in swabs collected from wounds pre-,intra- and postoperatively (7 days after surgery1). Change in bacterial load will be attributed to the effect of applying an antiseptic solution to wound dressings. | 7 days
  Wounds will be swabbed at end of surgery and then 7 days after surgery. Number and type of bacteria present will be analysed. Our hypothesis is that applying the antiseptic solution to the tie-over dressings will show a suppressed growth of bacteria when measured 7 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Saleh, MD, Principal Investigator — Department of Dermatology, Skåne University Hospital, Lund
Locations (1):
- Department of dermatology, Skåne university hospital, Lund, Sweden

REFERENCES:
- [Background] Saleh K, Sonesson A, Persson B, Riesbeck K, Schmidtchen A. A descriptive study of bacterial load of full-thickness surgical wounds in dermatologic surgery. Dermatol Surg. 2011 Jul;37(7):1014-22. doi: 10.1111/j.1524-4725.2011.02040.x. Epub 2011 May 25. PMID 21615603